CLINICAL TRIAL: NCT00990288
Title: The Role of a Topical Hemostatic Agent in Reducing Blood Loss in Unilateral Total Knee Arthroplasty
Brief Title: The Use of FLOSEAL to Reduce Bleeding in Total Knee Replacement Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 26078
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Blood Loss
Keywords: To decrease blood loss during knee surgery
MeSH Terms: conditions — Hemorrhage | interventions — FloSeal Matrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hemostatic Matrix (Experimental): 2 vials of Floseal applied once at the end of surgery
  Interventions: Drug: Hemostatic Matrix
- Control (No Intervention): No intervention.

INTERVENTIONS:
Drug: Hemostatic Matrix — FloSeal will be administered following the cementing of all knee components. Prior to release of the tourniquet and after the cement has cured, it will be applied to cut, exposed bone ends as well as the intra-articular soft tissues by the use of a delivery syringe, Direct manual pressure with a gauze sponge will be applied following its application for 2 minutes, ensuring that it adheres to the bleeding bone surface.
  Other Names: "FloSeal", a thrombin and collagen based agent
  Arms: Hemostatic Matrix

SUMMARY:
The purpose of this study is to determine if the agent, Floseal, can decrease the amount of blood patients lose after total knee replacement (TKR) surgery. If this product can be found to have an effect on bleeding, it may potentially reduce the problems associated with bleeding after knee replacement surgery such as pain, stiffness, and the need to have a blood transfusion. The subject's overall participation will be over a period of 6 weeks.

DETAILED DESCRIPTION:
This is a prospective double blind randomized clinical trial of patients requiring unilateral total knee arthroplasty. The patients will be randomized intra-operatively to receiving Floseal or no treatment.

Both the patient and the observers will be blinded to whether the subject received Floseal or no treatment. Only the operating surgeons will be aware of whether Floseal or no treatment was given.

As was performed in the pilot study, randomization of Floseal or no treatment will be performed using the sealed envelope technique. Randomization will occur at the time of surgery. The statistician is responsible for maintaining the randomization schedule and issuing the sealed envelopes. The inner envelope will contain whether Floseal or no treatment is to be given on a card which will be counter-signed by the surgeon at the time of surgery. The inner envelope will then be sealed, followed by sealing of the outer envelope. Following the procedure, the surgeon will then take the sealed and signed envelope to surgeon who will store and file it in a locked cabinet in his office. The patients study number will be on the outside surface of the envelopes.

ELIGIBILITY:
Inclusion Criteria:

* Single Knee replacement for arthritis of the knee

Exclusion Criteria:

* No inflammatory arthritis (ie. Rheumatoid arthritis)
* No allergies to cow meat (bovine allergies
* No history of bleeding disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2007-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Figgie, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion Criteria:
  1)Diagnosis of knee arthritis in patients medically suitable to undergo unilateral TKA.
  Pre-operative Exclusion Criteria:
  1. Known allergies to products of bovine origin.
  2. History of bleeding disorders.
  3. Pre- or peri-operative complication.
Period: Overall Study
Arm/Group | Hemostatic Matrix | Control
Started | 97 | 99
Completed | 97 | 99
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hemostatic Matrix | Control | Total
Number analyzed (Participants) | 97 | 99 | 196
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 73 | 93
  >=65 years | 77 | 26 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.78 (8.90) | 70.40 (10.47) | 71.58 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 71 | 136
  Male | 32 | 28 | 60
Region of Enrollment [Number; unit: participants]
  United States | 97 | 99 | 196

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin on Day 0 Compared to Preoperatively
Time Frame: preoperatively and on the day of surgery
Population: All patients enrolled in study were subject to analysis; occasionally a patient's levels were not taken or were not available for analysis for various reasons
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Hemostatic Matrix | Control
Number analyzed (Participants) | 96 | 98
g/dL | -1.277 (.880) | -1.241 (.883)

2. Primary Outcome: Change in Hemoglobin on Day 0 Compared to Preoperatively
Time Frame: preoperatively and day of surgery
Population: All patients enrolled in study were subject to analysis; occasionally a patient's levels were not taken or were not available for analysis.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Hemostatic Matrix | Control
Number analyzed (Participants) | 96 | 98
g/L | -4.484 (2.637) | -4.305 (2.682)

3. Primary Outcome: Change in Hemoglobin On Day 1 Compared to Preoperatively
Time Frame: preoperatively and one day after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Hemostatic Matrix | Control
Number analyzed (Participants) | 92 | 94
g/dL | -1.528 (1.132) | -1.816 (1.168)

4. Secondary Outcome: Range of Motion on Day 3
Time Frame: 3days postoperatively
Population: Patients whose range of motion at 3 day followup appointment was taken were included in analysis.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Hemostatic Matrix | Control
Number analyzed (Participants) | 97 | 97
degrees | 67.88 (14.54) | 68.96 (16.01)

5. Secondary Outcome: Visual Analog Pain Scale on Day 3
Description: A VAS is a measurement instrument that tries to measure a characteristic or attitude that cannot easily be measured.
  The pain VAS scale measures pain intensity on a scale of 0 to 10, with 0=no pain. A higher score indicates greater pain intensity.
Time Frame: 3 days postoperatively
Population: All patients whose pain score was collected were included in analysis.
Measure: Mean (Standard Deviation); unit: points on visual analog pain scale
Arm/Group | Hemostatic Matrix | Control
Number analyzed (Participants) | 96 | 98
points on visual analog pain scale | 2.99 (2.311) | 2.78 (2.44)

6. Primary Outcome: Change in Hematocrit on Day 1 Compared to Preoperatively
Time Frame: preoperatively and 1 day after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Hemostatic Matrix | Control
Number analyzed (Participants) | 92 | 94
g/L | -5.075 (3.298) | -5.749 (3.652)

7. Secondary Outcome: Range of Motion at Six Weeks
Time Frame: 6 weeks postoperatively
Population: Patients whose range of motion at 6-week followup appointment was taken were included in analysis.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Hemostatic Matrix | Control
Number analyzed (Participants) | 83 | 86
degrees | 111.41 (14.25) | 112.97 (12.92)

8. Primary Outcome: Change in Hemoglobin on Day 2 Compared to Preoperatively
Time Frame: preoperatively and two days after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Hemostatic Matrix | Control
Number analyzed (Participants) | 95 | 98
g/dL | -2.265 (1.443) | -2.359 (1.246)

9. Primary Outcome: Change in Hematocrit on Day 2 Compared to Preoperatively
Time Frame: preoperatively and two days after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Hemostatic Matrix | Control
Number analyzed (Participants) | 95 | 98
g/L | -7.013 (4.183) | -7.418 (3.904)

10. Primary Outcome: Drain Output
Time Frame: 24 hours postoperatively
Population: Drain output at 24 hours was recorded for all patients.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Hemostatic Matrix | Control
Number analyzed (Participants) | 97 | 99
mL | 711 (287) | 702 (314.7)

11. Primary Outcome: Autologous Amount of Transfusion
Time Frame: three days postoperatively
Measure: Mean (Standard Deviation); unit: units of blood
Arm/Group | Hemostatic Matrix | Control
Number analyzed (Participants) | 93 | 96
units of blood | .828 (.746) | .854 (.754)

12. Primary Outcome: Homologous Amount of Transfusion
Time Frame: three days postoperatively
Measure: Mean (Standard Deviation); unit: units of blood
Arm/Group | Hemostatic Matrix | Control
Number analyzed (Participants) | 95 | 95
units of blood | .247 (.525) | .337 (.738)

13. Secondary Outcome: Visual Analog Pain Scale at 6 Weeks
Description: as for outcome 5
Time Frame: 6 weeks postoperatively
Population: Patients whose pain level at 6-week followup appointment was taken were included in analysis.
Measure: Mean (Standard Deviation); unit: points on visual analog pain scale
Arm/Group | Hemostatic Matrix | Control
Number analyzed (Participants) | 90 | 88
points on visual analog pain scale | 2.753 (2.09) | 2.91 (2.17)

ADVERSE EVENTS:
Arm/Group | Hemostatic Matrix | Control
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/99
Other Adverse Events (participants affected / at risk) | 5/97 | 6/99
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hemostatic Matrix (N=97) | Control (N=99)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Deep Venous Thromboses (Vascular disorders) | 1 (1) | 1 (1)
Suture Abscess with Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Manipulation Under Anesthesia Needed to Achieve Improved Range of Motion (Surgical and medical procedures) | 2 (2) | 2 (2)
Paralytic Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes